CLINICAL TRIAL: NCT06578052
Title: Irinotecan Liposome in Combination With Capecitabine as Second-line Treatment for Advanced Pancreatic Cancer: Phase II Clinical Study
Brief Title: Irinotecan Liposome in Combination With Capecitabine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Junjie Hang (Other)
Responsible Party: Sponsor-Investigator, Junjie Hang, Associate chief physician, Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center
Organization: Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YW 2024-43
Record Dates: First submitted 2024-08-23; First posted 2024-08-29 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-08

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: "Irinotecan liposome: intravenous infusion, day 1, every 2 weeks (Q2W). Capecitabine: oral, twice daily (bid), days 1 to 7, take for one week and then have a one-week interval.
  Each 2-week period is considered a treatment cycle, with an expected treatment of 6 cycles. Subsequent maintenance treatment will be determined by the investigator's protocol until disease progression or intolerable toxicity occurs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Irinotecan liposome Capecitabine (Other): Irinotecan liposome: intravenous infusion, day 1, every 2 weeks (Q2W). Capecitabine: oral, twice daily (bid), days 1 to 7, take for one week and then have a one-week interval.
  Each 2-week period is considered a treatment cycle, with an expected treatment of 6 cycles. Subsequent maintenance treatment will be determined by the investigator's protocol until disease progression or intolerable toxicity occurs."
  Interventions: Drug: Irinotecan liposome Capecitabine

INTERVENTIONS:
Drug: Irinotecan liposome Capecitabine — Irinotecan liposome: intravenous infusion, day 1, every 2 weeks Capecitabine: oral, twice daily (bid), days 1 to 7, take for one week and then have a one-week interval.
  Each 2-week period is considered a treatment cycle, with an expected treatment of 6 cycles. Subsequent maintenance treatment will be determined by the investigator's protocol until disease progression or intolerable toxicity occurs."

SUMMARY:
Pancreatic cancer is a group of malignant tumors mainly originated from pancreatic ductal epithelium and follicular cells, with high degree of malignancy, insidious onset, difficult early diagnosis, rapid progression, short survival time, and one of the malignant tumors with the worst prognosis, which is known as the "king of cancers". In recent years, the incidence rate of pancreatic cancer has been increasing both at home and abroad. At present, the palliative treatment of advanced pancreatic cancer is still mainly based on chemotherapy, such as FOLFIRINOX regimen. And after standard first-line treatment, most of the patients have problems such as poor physical status, no standard treatment options and limited options available.

Capecitabine is a selective fluorouracil methionine salt antitumor drug, belongs to the pyrimidine class of antimetabolites, and is the precursor drug of 5-fluorouracil. Its first-line monotherapy for pancreatic cancer is 24% effective, and it is directly recommended by NCCN 2024 V2.0 as a second-line treatment for patients with pancreatic cancer who have failed gemcitabine therapy.The 2024 CSCO Guidelines for Pancreatic Cancer recommend the use of 5-fluorouracil (5-FU)-like regimens as a second-line treatment for patients who have been treated with a gemcitabine-based regimen as first-line treatment. In a clinical study exploring capecitabine in gemcitabine-treated patients with metastatic or unresectable locally advanced pancreatic cancer, 42 patients received oral capecitabine 1,250 mg/m2 twice daily (2,500 mg/m2/d) as intermittent therapy in 3-week cycles consisting of 2 weeks of dosing followed by 1 week of withdrawal. A total of 4 remissions were achieved in 42 evaluable patients, for an overall remission rate of 9.5%.

Irinotecan Hydrochloride Liposome Injection, the first domestic generic product developed by Shiyao Group, was launched in China in September 2023 with an approved indication for use in combination with 5-FU and calcium folinate (LV) in patients with metastatic pancreatic cancer that has progressed after treatment with gemcitabine. Liposomal irinotecan hydrochloride has been studied in a number of indications including biliary tract cancer, colorectal cancer, glioma, gastric cancer, small cell lung cancer, cervical cancer, breast cancer, head and neck cancer, esophageal cancer, and neuroendocrine cancer. In the bioequivalence trial of Shiyi Group's irinotecan hydrochloride liposome injection, the ORR rate reached 12.9%, the median PFS was 6.24 months, and the median OS was 10.38 months; indicating similar efficacy and a similar safety profile. A randomized, open-label, phase 3 NAPOLI 3 study and the first phase 3 trial comparing two combination chemotherapy regimens in the first-line treatment of patients with pancreatic ductal carcinoma head-to-head was designed to compare the efficacy and safety differences between the NALIRIFOX regimen (irinotecan liposomal, fluorouracil, and calcium folinic acid in combination with oxaliplatin) versus the doublet regimen (gemcitabine + albumin-conjugated paclitaxel) in the first-line treatment of metastatic pancreatic ductal carcinoma efficacy and safety differences in the treatment of metastatic pancreatic ductal cancer. The results showed that the median OS in the NALIRIFOX treatment group was 11.1 months, while the median OS in the dual combination treatment group was 9.2 months (HR=0.83; 95% CI 0.70-0.99; p=0.036).

Based on the above literature research, combined with the efficacy and safety advantages of irinotecan liposome chemotherapy combination regimen in patients with metastatic pancreatic cancer, we propose to carry out a phase II clinical study of irinotecan liposome combined with capecitabine in the second-line treatment of advanced pancreatic cancer. The aim is to explore the efficacy and safety of irinotecan liposomal chemotherapy combined with capecitabine in second-line unresectable or metastatic pancreatic cancer patients, and to explore more effective clinical options for patients with pancreatic cancer that has progressed after previous treatment.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, single-arm phase II study. It is expected to include 20 patients with unresectable/metastatic pancreatic cancer who have relapsed after standard treatment, and they will be treated with a regimen of liposomal irinotecan combined with capecitabine. The main research unit is the Shenzhen Hospital of the Chinese Academy of Medical Sciences Cancer Hospital. The study includes a screening period (within 28 days), a treatment period (an estimated 6 cycles, until disease progression or intolerable toxicity occurs), and a follow-up period (12 months for safety follow-up and progression-free survival (PFS) follow-up). Participants sign an informed consent form and undergo baseline examinations during the screening period. Patients who meet the inclusion and exclusion criteria enter the treatment period, and all participants complete the relevant examinations stipulated by the protocol during the treatment process to observe safety, tolerability, and efficacy. The same participant will only receive one dosing plan during the study period. After the end of the treatment period, the follow-up period begins

ELIGIBILITY:
Inclusion Criteria:

1. patients were fully aware of the study, participated voluntarily and signed the informed consent form (ICF);
2. aged ≥18 years and ≤80 years;
3. patients with histopathologically confirmed unresectable/metastatic pancreatic cancer;
4. imaging-confirmed tumor progression after prior treatment with a standard first-line regimen;
5. patients with at least one measurable target lesion according to RECIST 1.1 criteria;
6. Eastern Cooperative Oncology Group (ECOG) physical status score: 0-2;
7. expected survival time ≥ 3 months;
8. absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L, platelets ≥ 100 x 10^9/L and hemoglobin ≥ 90 g/L (not transfused with blood, blood products, or corrected with granulocyte colony-stimulating factor or other hematopoietic-stimulating factor in the 14 days prior to the laboratory test);
9. Liver and kidney function: serum creatinine ≤1.5 times the upper limit of normal value; AST and ALT ≤2.5 times the upper limit of normal value.

Liver and kidney function: serum creatinine ≤1.5 times the upper limit of normal value; AST and ALT ≤2.5 times the upper limit of normal value (≤5 times the upper limit of normal value for patients with liver metastases); total bilirubin ≤1.5 times the upper limit of normal value (≤3 times the upper limit of normal value for patients with liver metastases); 10. Women of childbearing potential must have had a negative pregnancy test (serum) within 7 days prior to enrollment and be willing to use an appropriate method of contraception for the duration of the trial and for 6 months after the last administration of the test drug.

-

Exclusion Criteria:

1. hypersensitivity to any of the study drugs or their components;
2. concomitant serious uncontrolled concurrent infections or other serious uncontrolled concomitant diseases, moderate or severe renal impairment; (e.g., progressive infections, uncontrollable hypertension, diabetes mellitus, etc.);
3. cardiac function and disease consistent with one of the following conditions

   1. Long QTc syndrome or QTc interval >480 ms;
   2. Complete left bundle branch block, degree II or degree III atrioventricular block;
   3. Severe, uncontrolled arrhythmia requiring pharmacologic therapy;
   4. New York Society of Cardiology classification ≥ grade III;
   5. Cardiac ejection fraction (LVEF) less than 50%;
   6. History of myocardial infarction, unstable angina, severe unstable ventricular arrhythmia or any other arrhythmia requiring treatment, history of clinically significant pericardial disease, or electrocardiographic evidence of acute ischemic or active conduction system abnormality within 6 months prior to recruitment.
4. active hepatitis B or C infection (hepatitis B virus surface antigen positive and hepatitis B virus DNA greater than 1x103 copies/mL; hepatitis C virus RNA greater than 1x103 copies/mL), except for asymptomatic chronic hepatitis B or hepatitis C carriers;
5. human immunodeficiency virus (HIV) infection (HIV-positive);
6. imaging confirmation of intestinal obstruction;
7. previous or current concurrent other malignancies (except effectively controlled non-melanoma basal cell carcinoma of the skin, carcinoma in situ of the breast/cervix, and other malignancies that have been effectively controlled without treatment within the past five years);
8. pregnant and lactating women and patients of childbearing age who do not wish to use contraception;
9. patients with other malignant tumors requiring treatment;
10. patients who, in the judgment of the investigator, are not suitable for participation in this study.
11. history of pulmonary hemorrhage/coughing up ≥ grade 2 (defined as at least 2.5 mL of bright red blood) within 1 month prior to the first dose of drug;
12. a predisposition to arterial embolism, severe hemorrhage (other than bleeding due to surgery), and severe bleeding within 6 months prior to first dose;
13. a combination of symptomatic brain metastases, meningeal metastases, spinal cord tumor invasion, and spinal cord compression
14. use of strong inhibitors or inducers of CYP3A4, CYP2C8, and UGT1A1 within 14 days prior to receiving study drug therapy
15. who have used other clinical trial medications within 1 month prior to the first dose;
16. pregnant or lactating female patients, subjects of childbearing age who refuse to accept contraception; -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | TFrom date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Progression-Free Survival (PFS)

SECONDARY OUTCOMES:
Objective Response Rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Objective Response Rate (ORR)
Disease Control Rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Disease Control Rate (DCR)
Overall Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Overall Survival (OS)

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No